

## MAKERERE UNIVERSITY COLLEGE OF HEALTH SCIENCES UNIVERSITY OF CALIFORNIA, SAN FRANCISCO

## INFORMED CONSENT TO PARTICIPATE IN A RESEARCH STUDY

## ASSESSMENT OF VITAL STATUS AND OTHER MEDICAL HISTORY FOR THE XPEL TB STUDY

I am working with a research team at Makerere University College of Health Sciences. I was looking for you because you were evaluated for tuberculosis (TB) at [CLINIC NAME] about six months ago. Are you available to talk for a few minutes?

I would like to invite you to participate in a survey, which includes questions about TB-related evaluation or treatment you have had since your visit to [CLINIC NAME]. I would also like to ask you about your HIV status and, if you are HIV-infected, when you started ART. This survey should take about 5-10 minutes. You can ask questions, refuse to answer specific questions or stop the survey at any time. There is a risk that participating in this survey could result in disclosure of your personal medical information, including HIV and TB status. However, we have strong protections in place to minimize this risk. Your responses to these questions will be stored in a secure location at [CLINIC NAME] before being transported to Kampala by a member of the study team for secure storage in our study office and entry into a passwordprotected database. Data shared with other researchers for analysis will exclude all information that could be used to identify you. In addition, if this study is published or presented somewhere, names and other information that might identify you will not be used.

Participating in this survey is voluntary. You have the right to decline or withdraw your participation at any time. You will not be charged any costs for participating nor will you receive compensation for your time.

If you have any concerns or questions about this study at any time, you can contact the Principal Investigator in Uganda, Dr. Achilles Katamba, at 256-753-040-922. You may also contact the Chairperson of the Research Ethics Committee at the School of Public Health Makerere University, Dr. Suzanne Kiwanuka, at +256772963074/ +256704663074 for questions concerning your rights while you participate in the survey.

This study is funded by the National Institutes of Health (NIH) through the University of California, San Francisco (UCSF).

Do you have any questions or concerns about the study?

## **PARTICIPANT**



IRB NUMBER: 17-21505 IRB APPROVAL DATE: 04/22/2020 IRB EXPIRATION DATE: 04/21/2021

You have been offered a copy of this consent form to keep. PARTICIPATION IN RESEARCH IS VOLUNTARY. You have the right to decline to participate or to withdraw at any point in this study without penalty or loss of benefits to which you are otherwise entitled. If you wish to participate in this study, please sign below.

| Date | Participant's Signature or Mark |
|---|---|
| (Do not date here if participant cannot re | ad and write) |
| Date | Signature of Witness Attending Consent |
| HEALTH WORKER | |
| Date | Signature of Person Obtaining Consent |

